CLINICAL TRIAL: NCT04466384
Title: Bispectral Index and Levels of Sedation With Propofol With/Without Remifentanil in Healthy Volunteers (SONORA)
Acronym: SONORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MDT19049SONORA
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: The subjects will receive two regimens of anesthesia with different drug combinations, with at least a 1-week washout period between regimens. Subjects will be sequentially assigned to start with either propofol or propofol with remifentanil regiments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Propofol (Other): Subjects will be sequentially assigned to start with propofol or propofol with remifentanil. Propofol will be started at a concentration of 0.5 µg/ml followed by incremental increases in the target effect-site concentrations of 1.5, 2, 2.5, 3, 4, 6, and 8 µg/ml until a MOAA/S score less than 2 is reached.
  Interventions: Device: BIS
- Propofol with Remifentanil (Other): Subjects will be sequentially assigned to start with propofol or propofol with remifentanil. Approximately 2 minutes before starting propofol, to attain an effect-site targeted concentration of remifentanil of 4 ng/ml, remifentanil will be given by a continuous infusion. Within approximately 7 minutes, the infusion rate of Remifentanil may be adjusted to maintain the effect-site concentration of remifentanil of 4 ng/ml throughout the study.
  Interventions: Device: BIS

INTERVENTIONS:
Device: BIS — Subjects will be sequentially assigned to the propofol or propofol and remifentanil group. The purpose is to capture the BIS value in association with these anesthetics.

SUMMARY:
The purpose of this study is investigate the relationship between BIS™ and propofol with/without remifentanil across a wide range of hypnotic states.

DETAILED DESCRIPTION:
This is a single-center, prospective, non-randomized, cross-over study to collect data to evaluate the relationship between BIS™ and anesthetic regimens. The subjects will receive two regimens of anesthesia with different drug combinations, with at least a 1-week washout period between regimens. Subjects will be sequentially assigned to start with either Propofol (P) or Propofol with 4 ng/ml of Remifentanil (R) regimens while BIS™ bilateral sensor placed on the subject's forehead. The Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scale, refer to Appendix A, will be used to measure the level of alertness in sedated subjects with Tetanic Electrical Stimulation (TES) being used once subjects reach a MOAA/S score <2.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (ASA physical status 1), male or female subjects between the ages of 18 to 60 years;
2. Completion of a health screening for a medical history by a licensed physician, nurse practitioner or physician assistant;
3. Vital signs must be within the following ranges to be included: Vital signs measured sitting after 3 minutes rest; heart rate: 45-90 bpm; systolic blood pressure: 110-140; diastolic blood pressure: 50-90. Out-of-range vital signs may be repeated once. [Pre-dose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) before study drug administration. The Principal Investigator or designee will verify the eligibility of each subject before dosing];

Exclusion Criteria:

1. Has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes, or other medical sensors [self-reported];
2. Known neurological disorder (e.g., epilepsy, the presence of a brain tumor, a history of brain surgery, hydrocephalic disorders, depression needing treatment with anti-depressive drugs, a history of brain trauma) [self-reported and assessment by PI or delegate];
3. Known cardiovascular disease (e.g., hypertension, coronary artery disease, prior acute myocardial infarction, any valvular and/or myocardial disease involving a decrease in ejection fraction, arrhythmias, which are either symptomatic or require continuous medication/ pacemaker/ automatic internal cardioverter defibrillator), current implanted pacemaker or automatic internal cardioverter defibrillator [self-reported and assessment by PI or delegate];
4. Has a clinically significant abnormal finding on medical history, physical examination, clinical laboratory tests, or ECG at the screening [self-reported and assessment by PI or delegate];
5. Recent use of psychoactive medication (e.g., benzodiazepines, antiepileptic drugs, ADHD medication, Parkinson's medication, anti-depressant drugs, opioids) [self-reported and assessment by PI or delegate];
6. Subjects with known gastric diseases [self-reported and assessment by PI or delegate];
7. Has a positive urine cotinine test or urine drug screen or oral ethanol test [POC testing];
8. Known history of allergic or adverse response to drugs to be administered [self-reported];
9. Known history of complications relating to previous general anesthesia or conscious sedation [self-reported and assessment by PI or delegate];
10. Known history of malignant hyperthermia [self-reported and assessment by PI or delegate];
11. Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate];
12. Has a clinically significant abnormal ECG [assessment by PI or delegate];
13. Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate];
14. Pregnant or lactating women [assessed by urine test and self-reported];
15. Subjects with tattooed skin specific to the sensor placement areas (forehead, fingers, chest) [self-reported and assessment by PI or delegate];
16. The subject must not take any prescription medication, except female hormonal contraceptives or hormone replacement therapy, from 146 days before the dosing until the end-of-study visit without evaluation and approval by the Investigator. Subjects who participated in a previous clinical trial who received a required FDA approved concomitant medication, for example, naltrexone, but were not randomized may be considered for participation in this study if they meet the washout requirement [assessment by PI or delegate];

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited healthy, non-smoking (or has refrained from smoking for 2 days) subjects, 18 to 60 years of age. The subjects were distributed across both sexes as equally as practical.
Pre-assignment Details: During the study, 34 subjects were consented. 6 subjects were inclusion / exclusion criteria screen failures after consent leaving 28 enrolled subjects. Of these 28 enrolled subjects, 4 subjects were withdrawn due to safety events leaving 24 subjects to be assigned to randomization arms.
Groups:
- Propofol First: Participants first received two regimens of Propofol (first phase). After a 1-week washout period, then received two regimens of Propofol with 4 ng/ml Remifentanil (cross over phase).
- First Propofol With Remifentanil: Participants first received two regimens of Propofol with 4 ng/ml Remifentanil (first phase). After a 1-week washout period, then received two regimens of Propofol (cross over phase).
Period: First Phase
Arm/Group | Propofol First | First Propofol With Remifentanil
Started | 14 | 10
Completed | 12 | 10
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Missing data | 1 | 0
Period: Cross Over Phase
Arm/Group | Propofol First | First Propofol With Remifentanil
Started | 14 | 10
Completed | 13 | 9
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: the subjects received two regimens of anesthesia with different drug combinations, with at least a 1-week washout period between regimens. Once the pre-procedure part was completed, the subject was sequentially assigned to start with either Propofol (P) or Propofol with 4 ng/ml of Remifentanil (R) regimens.
  The Safety Population includes all ITT subjects (results will be shown accordingly).
Groups:
- Randomized Study Participants: Baseline measures are reported for subjects who were enrolled and randomized to Propofol first or First Propofol with Remifentanil arms (n=24). Baseline measurements are not reported for subjects who were screen failures (n=6) or withdrawn due to safety events (n=4).
Arm/Group | Randomized Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24
Skin Pigmentation [Number; unit: participants] — The Fitzpatrick scale was used to evaluate skin pigmentation
  participants
    Very Light | 7
    Olive Hue | 4
    Dark Olive | 3
    Extremely Dark | 10

OUTCOME MEASURES:

1. Primary Outcome: BIS50
Description: To determine BIS50 (BIS™ value at which 50% of patients will be unresponsive at given drug concentrations) and other dose-response parameters. BIS™ is a scale 0-100 with values near 100 represent an "awake" clinical state while 0 denotes the maximal EEG effect possible (i.e., an isoelectric EEG). Responsiveness is measured using the Modified Observer's Assessment of Alertness/ Sedation (MOAA/S). Below a MOAA/S of 2, responsiveness is measured with Tetanic Electrical Stimulation (TES). The subject will receive one stimulation of 50mA, 50 Hz for 5 seconds. Their response, such as withdrawal of the extremity, a facial grimace, or a verbal groan will be recorded. Approximately 2 minutes after this assessment, the BIS™ value will be recorded. When the subject does not respond to the TES stimulation, they will be considered unresponsive and that BIS™ value will be used to determine the BIS50.
Time Frame: 4 hours
Population: Intention to Treat (ITT)
Measure: Number (95% Confidence Interval); unit: BIS50 Index Score
Arm/Group | Propofol | Propofol With Remifentanil
Number analyzed (Participants) | 24 | 24
BIS50 Index Score | 60.4 [57.7 to 63.0] | 71.6 [69.0 to 74.6]

2. Secondary Outcome: BIS95
Description: To determine BIS95 (BIS™ value at which 95% of patients will be unresponsive at given drug concentrations) and other dose-response parameters. BIS™ is a scale 0-100 with values near 100 represent an "awake" clinical state while 0 denotes the maximal EEG effect possible (i.e., an isoelectric EEG). Responsiveness is measured using the Modified Observer's Assessment of Alertness/Sedation (MOAA/S). Below a MOAA/S of 2, responsiveness is measured with Tetanic Electrical Stimulation (TES). The subject will receive one stimulation of 50mA, 50 Hz for 5 seconds. Their response, such as withdrawal of the extremity, a facial grimace, or a verbal groan will be recorded. Approximately 2 minutes after this assessment, the BIS™ value will be recorded. When the subject does not respond to the TES stimulation, they will be considered unresponsive and that BIS™ value will be used to determine the BIS95.
Time Frame: 4 hours
Population: Intention to Treat (ITT)
Measure: Number (95% Confidence Interval); unit: BIS95 index score
Arm/Group | Propofol | Propofol With Remifentanil
Number analyzed (Participants) | 24 | 24
BIS95 index score | 47.7 [40.5 to 51.7] | 63.1 [57.3 to 66.2]

ADVERSE EVENTS:
Time Frame: 48 hours
Description: For the adverse event analysis, events were analyzed for the two treatment groups (Propofol + Opioid vs. Propofol).
Groups:
- Propofol First (First Phase); Propofol First (Cross Over Phase): Participants first received two regimens of Propofol (first phase). After a 1-week washout period, then received two regimens of Propofol with 4 ng/ml Remifentanil (cross over phase).
- First Propofol With Remifentanil (First Phase); First Propofol With Remifentanil (Cross Over Phase): Participants first received two regimens of Propofol with 4 ng/ml Remifentanil (first phase). After a 1-week washout period, then received two regimens of Propofol (cross over phase).
Arm/Group | Propofol First (First Phase) | First Propofol With Remifentanil (First Phase) | Propofol First (Cross Over Phase) | First Propofol With Remifentanil (Cross Over Phase)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10 | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 0/14 | 3/10 | 8/14 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol First (First Phase) (N=14) | First Propofol With Remifentanil (First Phase) (N=10) | Propofol First (Cross Over Phase) (N=14) | First Propofol With Remifentanil (Cross Over Phase) (N=10)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
While there are known risks with providing general anesthesia to adults, this study was deemed to be a non-significant risk study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT04466384/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT04466384/SAP_004.pdf